CLINICAL TRIAL: NCT05409378
Title: HLT® Meridian® TAVR Valve System Early Feasibility Study for Aortic Regurgitation
Acronym: RIVAL - AR EFS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: HLT Business Decision
Sponsor: HLT Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLT2101
Record Dates: First submitted 2022-05-24; First posted 2022-06-08 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Aortic Regurgitation
Keywords: Aortic Valve; Regurgitation; Transcatheter; Replacement
MeSH Terms: conditions — Aortic Valve Insufficiency; Gastroesophageal Reflux | interventions — Meridians

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- The HLT® Meridian® TAVR Valve (Experimental): Transcatheter aortic valve replacement with the HLT Meridian TAVR Valve
  Interventions: Device: The HLT® Meridian® TAVR Valve (Meridian® with TriVentTM Anticalcification Treatment Valve and Pathfinder® Delivery System)

INTERVENTIONS:
Device: The HLT® Meridian® TAVR Valve (Meridian® with TriVentTM Anticalcification Treatment Valve and Pathfinder® Delivery System) — Aortic valve replacement with the HLT Meridian TAVR Valve to treat aortic regurgitation

SUMMARY:
To evaluate the safety and performance of The Meridian® TAVR Valve in patients with severe aortic regurgitation who present at high risk for aortic valve replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has evidence of severe aortic regurgitation as assessed by the independent echo core lab according to an integrative multiparametric based on ASE (American Society of Echocardiography) guidelines considering qualitative and quantitative measures.
2. Symptoms due to severe aortic regurgitation with a NYHA Functional Classification of II or greater
3. Documented aortic valve annular diameter ≥ 21 and ≤ 26 mm (associated perimeter range is 66.0 - 81.7 mm or associated area range of 346 - 531 mm^2) measured by the MSCT Core Lab assessment of pre-procedure imaging
4. Documented heart team agreement of high risk for surgical aortic valve replacement (SAVR)
5. Geographically available, willing to comply with follow-up and able to provide written informed consent.

Exclusion Criteria:

1. Congenital, unicuspid or bicuspid aortic valve which could compromise procedural success
2. Severe mitral or tricuspid valve regurgitation
3. Moderate to severe mitral stenosis
4. Myocardial infarction within the past 30 days*
5. Echocardiographic evidence of intracardiac mass, thrombus or vegetation
6. Left Ventricular Ejection Fraction (LVEF) < 35%
7. Severe pulmonary hypertension with pulmonary systolic pressure greater than two-thirds of systemic pressure
8. Hemodynamic instability requiring inotropic drug therapy within the past 30 days
9. Untreated clinically significant coronary artery disease requiring revascularization
10. Any therapeutic invasive cardiac procedure performed or planned to perform within 30 days of the index procedure, except for PCI which is performed within 7 days prior to the index procedure*
11. Presence of significant aortic disease such as atheroma, thrombus, dissection (> 50 mm in diameter or which could be considered high risk for dissection) or aneurysm which precludes safe implant delivery
12. Blood dyscrasias defined as leukopenia (White blood cell count < 1,000 cell/mm^3), anemia (hemoglobin < 9.0 g/dL), thrombocytopenia (platelet count < 50,000 cells/mm^3), history of bleeding diathesis or coagulopathy
13. Patient ineligible for or refuses blood transfusions
14. Unfavorable peripheral vascular anatomy or disease (e.g. severe obstructive calcification, severe tortuosity) that would preclude passage of 18F catheters from the femoral arterial access to the aorta by the MSCT Core Lab assessment of pre-procedure imaging
15. Active peptic ulcer or gastrointestinal bleeding requiring hospitalization or transfusion within the past 90 days, that would not allow treatment with the protocol antiplatelet regimen post implant *
16. Symptoms of carotid or vertebral artery disease (e.g. stroke or transient ischemic attack) within past 6 months, or treatment of carotid stenosis within past two months*

    * At the time of procedure, if a subject's medical status has changed since enrollment, the subject shall be re-evaluated for eligibility

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Mortality at 30 days | 30-Days
  The primary safety endpoint is all-cause mortality at 30 days

SECONDARY OUTCOMES:
Technical Success - A composite endpoint per VARC-3, defined as meeting the following: | Immediately after procedure
  * Freedom from Mortality
  * Successful access, delivery of the device, and retrieval of the delivery system
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complication
Device Success- A composite endpoint per VARC-3, defined as meeting the following: | 30 Days
  * Technical Success
  * Freedom from mortality
  * Freedom from surgery or intervention related to the device a or to a major vascular or access-related or cardiac structural complication
  * Intended performance of the valve (mean gradient < 20 mmHg, peak velocity < 3 m/s, Doppler velocity index ≥ 0.25, and less than moderate aortic regurgitation.
Post-procedural Valve Performance - EOA assessed via Echo | Discharge (or day 7), 30 days, 6, 12, 24, 36, 48 and 60 months
  • Aortic valve effective orifice area (EOA; cm^2)
Post-procedural Valve Performance- Aortic Regurgitation (AR) assessed via Echo | Discharge (or day 7), 30 days, 6, 12, 24, 36, 48 and 60 months
  • Severity of aortic valve regurgitation (AR; graded scale)
Post-procedural Valve Performance - Aortic Valve Gradient assessed via Echo | Discharge (or day 7), 30 days, 6, 12, 24, 36, 48 and 60 months
  • Aortic valve gradient (mean and peak; mmHg)
Adverse Events | Up to 5 years following enrollment
  All adverse events will be assessed throughout the five (5) year follow up period per VARC-3 definitions

CONTACTS AND LOCATIONS:
Overall Officials: Kendra Grubb, MD, Principal Investigator — Emory University; Charles Davidson, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - The Christ Hospital, Cincinnati, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No